CLINICAL TRIAL: NCT03662100
Title: A Safety, Tolerability, and Pharmacokinetic Study of Injections of LY3074828 Solution Using Investigational 1-mL Pre-filled Syringes and Investigational 2-mL Autoinjector in Healthy Subjects
Brief Title: A Study of Two Formulations of LY3074828 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16618; I6T-MC-AMAR (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Results first posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-05-01

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (6):
- Test 1: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-milligram/milliliter [mg/mL]) administered subcutaneously (SC) via an auto-injector (AI) in arm.
  Interventions: Biological: LY3074828; Device: Auto-injector (AI)
- Test 2: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in thigh.
  Interventions: Biological: LY3074828; Device: Auto-injector (AI)
- Test 3: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in abdomen.
  Interventions: Biological: LY3074828; Device: Auto-injector (AI)
- Reference 1: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in pre-filled syringe (PFS) administered as subcutaneous (SC) injection in arm.
  The second injection was administered 20 (±2) minutes after the first injection.
  Interventions: Drug: LY3074828; Device: Prefilled syringe (PFS)
- Reference 2: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in thigh.
  The second injection was administered 20 (±2) minutes after the first injection.
  Interventions: Drug: LY3074828; Device: Prefilled syringe (PFS)
- Reference 3: 250 mg LY3074828 (Experimental): Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in abdomen.
  The second injection was administered 20 (±2) minutes after the first injection.
  Interventions: Drug: LY3074828; Device: Prefilled syringe (PFS)

INTERVENTIONS:
Biological: LY3074828 — Administered SC
  Arms: Test 1: 250 mg LY3074828; Test 2: 250 mg LY3074828; Test 3: 250 mg LY3074828
Drug: LY3074828 — Administered SC
  Arms: Reference 1: 250 mg LY3074828; Reference 2: 250 mg LY3074828; Reference 3: 250 mg LY3074828
Device: Auto-injector (AI) — AI to administer LY3074828
  Arms: Test 1: 250 mg LY3074828; Test 2: 250 mg LY3074828; Test 3: 250 mg LY3074828
Device: Prefilled syringe (PFS) — PFS to administer LY3074828
  Arms: Reference 1: 250 mg LY3074828; Reference 2: 250 mg LY3074828; Reference 3: 250 mg LY3074828

SUMMARY:
The purpose of this study is to look at the amount of the study drug, LY3074828, that gets into the blood stream and how long it takes the body to get rid of LY3074828 when given as different formulations. The tolerability of LY3074828 will also be evaluated and information about any side effects experienced will be collected.

Screening is required within 28 days prior to the start of the study. For each participant, the study will last about 12 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria: Healthy participants.

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 8 weeks of screening, or intend to during the study
* Must not have been treated with steroids within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to Day 1
* Must not have significant allergies to humanised monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or severe post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-06 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Test 1: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-milligram/milliliter [mg/mL]) administered subcutaneously(SC) via an auto-injector (AI) in arm.
- Reference 1: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in pre-filled syringe (PFS) administered as subcutaneous (SC) injection in arm.The second injection was administered 20 (±2) minutes after the first injection.
- Reference 3: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in abdomen.The second injection was administered 20 (±2) minutes after the first injection.
Period: Overall Study
Arm/Group | Test 1: 250 mg LY3074828 | Test 2: 250 mg LY3074828 | Test 3: 250 mg LY3074828 | Reference 1: 250 mg LY3074828 | Reference 2: 250 mg LY3074828 | Reference 3: 250 mg LY3074828
Started | 11 | 11 | 11 | 11 | 11 | 11
Received at Least One Dose of Drug | 11 | 11 | 11 | 11 | 11 | 11
Completed | 11 | 11 | 11 | 11 | 11 | 11
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Test 1: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an auto-injector (AI) in arm.
- Reference 2: 250 mg LY3074828: Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in thigh.The second injection was administered 20 (±2) minutes after the first injection.
- Total: Total of all reporting groups
Arm/Group | Test 1: 250 mg LY3074828 | Test 2: 250 mg LY3074828 | Test 3: 250 mg LY3074828 | Reference 1: 250 mg LY3074828 | Reference 2: 250 mg LY3074828 | Reference 3: 250 mg LY3074828 | Total
Number analyzed (Participants) | 11 | 11 | 11 | 11 | 11 | 11 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (14.3) | 39.9 (13.7) | 45.4 (9.4) | 44.1 (14.7) | 42.8 (12.3) | 45.0 (12.9) | 43.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 6 | 6 | 7 | 7 | 39
  Male | 4 | 5 | 5 | 5 | 4 | 4 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 5 | 4 | 4 | 7 | 28
  Not Hispanic or Latino | 7 | 7 | 6 | 7 | 7 | 4 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 4 | 4 | 1 | 4 | 0 | 14
  White | 8 | 6 | 6 | 10 | 7 | 11 | 48
  More than one race | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 11 | 11 | 11 | 11 | 66

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3074828 by Device
Description: Pharmacokinetics: Cmax of LY3074828
Time Frame: Day 1: 0, 2, 6 hours (hr), Day 2: 24 hr, Day 4, Day 8, Day 11, Day 15, Day 22, Day 29, Day 43, Day 57, Day 71, Day 85, Post dose
Population: All participants who received at least one dose of study drug. Per protocol, PK analysis were performed to compare all PFS participants together versus all AI participants together.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Groups:
- 250 mg LY3074828 AI: Test 1: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an auto-injector (AI) in arm.
  Test 2: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in thigh.
  Test 3: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in abdomen.
- 250 mg LY3074828 PFS: Reference 1: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in pre-filled syringe (PFS) administered as subcutaneous (SC) injection in arm.
  Reference 2: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in thigh.
  Reference 3: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in abdomen.
  The second injection was administered 20 (±2) minutes after the first injection.
Arm/Group | 250 mg LY3074828 AI | 250 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
micrograms per milliliter (μg/mL) | 22.2 (40) | 18.7 (34)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Infinity (AUC(0-∞)) of LY3074828 by Device
Description: Pharmacokinetics: Area Under the Concentration versus Time Curve From Time Zero to Infinity (AUC(0-∞)) of LY3074828
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*day per millileter (μg*day/mL)
Arm/Group | 250 mg LY3074828 AI | 250 mg LY3074828 PFS
Number analyzed (Participants) | 33 | 33
microgram*day per millileter (μg*day/mL) | 357 (38) | 340 (38)

3. Primary Outcome: Visual Analogue Scale (VAS) Pain Assessment by Device
Description: The VAS is a single-item participant-rated assessment of injection pain. Score is reported on a continuous scale of 0 to 100. Higher values indicate more pain.
Time Frame: Day 1: 1, 5 (±1.5) and 15 (±2) minutes
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- 250 mg LY3074828 AI First Injection: Test 1: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an auto-injector (AI) in arm.
  Test 2: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in thigh.
  Test 3: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (1 x 2-mL 125-mg/mL) administered SC via an AI in abdomen.
- 250 mg LY3074828 PFS First Injection: Reference 1: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in pre-filled syringe (PFS) administered as subcutaneous (SC) injection in arm.
  Reference 2: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in thigh.
  Reference 3: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in abdomen.
- 250 mg LY3074828 PFS Second Injection: Reference 1: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in pre-filled syringe (PFS) administered as subcutaneous (SC) injection in arm.
  Reference 2: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in thigh.
  Reference 3: 250 mg LY3074828 Participants received 250 mg LY3074828 solution formulation (2 x 1-mL 125-mg/mL) in PFS administered as SC injection in abdomen.
  The second injection was administered 20 (±2) minutes after the first injection.
Arm/Group | 250 mg LY3074828 AI First Injection | 250 mg LY3074828 PFS First Injection | 250 mg LY3074828 PFS Second Injection
Number analyzed (Participants) | 33 | 33 | 33
millimeter
  1 min | 25.2 (20.0) | 22.6 (18.3) | 18.3 (15.1)
  5 min (±1.5) | 12.0 (15.8) | 6.1 (7.0) | 6.0 (6.7)
  15 min (±2) | 1.9 (3.1) | 2.4 (2.8) | 2.2 (4.3)

4. Primary Outcome: Visual Analogue Scale (VAS) Pain Assessment by Device and Injection Site Location
Description: as for outcome 3
Time Frame: Day 1: 1, 5 (±1.5) and 15 (±2) minutes
Population: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | 250 mg LY3074828 AI First Injection | 250 mg LY3074828 PFS First Injection | 250 mg LY3074828 PFS Second Injection
Number analyzed (Participants) | 33 | 33 | 33
millimeter
  Arm: 1 min: number analyzed (Participants) | 11 | 11 | 11
  Arm: 1 min | 25.9 (17.2) | 19.0 (12.0) | 15.6 (12.3)
  Arm: 5 min (±1.5): number analyzed (Participants) | 11 | 11 | 11
  Arm: 5 min (±1.5) | 5.6 (5.4) | 4.5 (5.5) | 5.0 (6.0)
  Arm: 15 min (±2): number analyzed (Participants) | 11 | 11 | 11
  Arm: 15 min (±2) | 2.6 (4.8) | 1.8 (2.4) | 2.0 (2.9)
  Thigh: 1 min: number analyzed (Participants) | 11 | 11 | 11
  Thigh: 1 min | 26.8 (15.5) | 19.6 (20.9) | 20.5 (19.6)
  Thigh: 5 min (±1.5): number analyzed (Participants) | 11 | 11 | 11
  Thigh: 5 min (±1.5) | 13.1 (12.3) | 6.2 (6.6) | 7.9 (7.8)
  Thigh:15 min (±2): number analyzed (Participants) | 11 | 11 | 11
  Thigh:15 min (±2) | 0.9 (1.3) | 3.0 (3.6) | 3.5 (6.7)
  Abdomen: 1 min: number analyzed (Participants) | 11 | 11 | 11
  Abdomen: 1 min | 22.9 (27.2) | 29.2 (20.6) | 18.7 (13.4)
  Abdomen: 5 min (±1.5): number analyzed (Participants) | 11 | 11 | 11
  Abdomen: 5 min (±1.5) | 17.4 (23.3) | 7.5 (8.8) | 5.0 (6.4)
  Abdomen: 15 min (±2): number analyzed (Participants) | 11 | 11 | 11
  Abdomen: 15 min (±2) | 2.2 (2.1) | 2.4 (2.4) | 1.2 (1.9)

ADVERSE EVENTS:
Time Frame: Up To 85 Days
Description: All participants who received at least one dose of study drug.
Arm/Group | Test 1: 250 mg LY3074828 | Test 2: 250 mg LY3074828 | Test 3: 250 mg LY3074828 | Reference 1: 250 mg LY3074828 | Reference 2: 250 mg LY3074828 | Reference 3: 250 mg LY3074828
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/11 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 3/11 | 6/11 | 2/11 | 3/11 | 6/11 | 4/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test 1: 250 mg LY3074828 (N=11) | Test 2: 250 mg LY3074828 (N=11) | Test 3: 250 mg LY3074828 (N=11) | Reference 1: 250 mg LY3074828 (N=11) | Reference 2: 250 mg LY3074828 (N=11) | Reference 3: 250 mg LY3074828 (N=11)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Refraction disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03662100/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/00/NCT03662100/SAP_001.pdf